CLINICAL TRIAL: NCT00032409
Title: The Effects of Music Therapy-Based Stress Reduction on Bone Marrow Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AT000895-01 (NIH)
Record Dates: First submitted 2002-03-20; First posted 2002-03-22 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Bone Marrow Transplantation; Stem Cell Transplantation
Keywords: Music Therapy; Relaxation Therapy; Stress Reduction; Bone Marrow Transplantation; Stem Cell Transplantation

INTERVENTIONS:
Behavioral: Music therapy-based relaxation/stress reduction

SUMMARY:
The purpose of this study is to determine the effects of music therapy-based relaxation stress/reduction strategies on the frequency/severity of toxic side-effects of marrow ablative chemotherapy and the timing of immune reconstitution in patients undergoing bone marrow/stem cell transplantation.

DETAILED DESCRIPTION:
The regimen-related toxicities associated with bone marrow transplantation (BMT) can be severe and even life threatening. The overall goal of this randomized controlled pilot study in BMT patients is to determine the effect of relaxation/stress reduction strategies on: (1) the frequency/severity of toxic side effects of marrow ablative chemotherapy, and (2) the timing of immune reconstitution. Substantial literature indicates that music therapy-based interventions are effective in inducing relaxation and also affect immune function by modulating circulating and salivary levels of such agents as cortisol, immunoglobulin A, interleukin-1, natural killer cells, and a variety of other immune system-related substances. Over the past two years, we have provided music therapy-based stress reduction/relaxation interventions to a convenience sample of patients undergoing BMT. Preliminary findings from this pilot feasibility study demonstrate that patients report significantly decreased pain (p< .004) and sense of nausea (p < .001) following an intervention. Average time-to-engraftment was 13.5 (+/- 2.85) days as compared to 15.5 (+/- 4.40) days (p < .O1) for a group of historical controls matched on diagnosis, type of transplant, conditioning regimen, date of transplant, age, and gender. Although highly promising, our data are limited by lack of randomization, an appropriate control condition, measurement of psychologic factors known to influence outcome in BMT, and systematic monitoring of early phase markers of immune reconstitution that could help explain the phenomena we have observed. This proposal corrects these shortcomings and especially highlights the potential mediational effect of cytokine release on regimen-related toxicities and the timing of immune reconstitution.

ELIGIBILITY:
Inclusion:

Recipient of bone marrow/stem cell transplant

Exclusion:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2001-08; Study Completion 2004-06

CONTACTS AND LOCATIONS:
Overall Officials: Olle Jane Z. Sahler, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States